CLINICAL TRIAL: NCT07120477
Title: Esketamine Versus Crisis Response Planning Versus Optimized Treatment as Usual for Suicide Prevention: A Pragmatic Controlled Trial in Two Brazilian Cities
Acronym: SAVE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rodolfo Furlan Damiano, Post-doc Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 89878225.0.0000.0068
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Suicide Prevention; Ketamine; Crisis Response Plan
Keywords: Suicide Prevention; Ketamine; Crisis Response Plan
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Esketamine plus optimized usual treatment (Experimental): Single esketamine infusion (0.5 mg/kg over 40 minutes) plus optimized usual treatment (early psychiatric follow-up within one week)
  Interventions: Drug: Intravenous Esketamine
- Crisis Response Planning plus Optimized Usual Treatment (Experimental): Crisis Response Planning intervention (structured safety planning) plus optimized usual treatment (early psychiatric follow-up within one week)
  Interventions: Other: Crisis Response Planning intervention (structures safety planning)
- Optimized Usual Treatment Only (Active Comparator): Optimized usual treatment alone (enhanced standard care with early psychiatric follow-up within one week)
  Interventions: Drug: Intravenous Esketamine; Other: Crisis Response Planning intervention (structures safety planning)

INTERVENTIONS:
Drug: Intravenous Esketamine — Single-session intravenous esketamine infusion (0.5 mg/kg) administered over 40 minutes in a medical setting with continuous monitoring of vital signs, blood pressure, ECG, and oxygen saturation for 4 hours post-infusion. Administration supervised by trained medical staff with emergency protocols available. Participants will be discharged 24 hours post-infusion if no clinical complications arise, with ambulatory evaluations at 48 hours, 72 hours, and 7 days post-infusion.
  Arms: Esketamine plus optimized usual treatment; Optimized Usual Treatment Only
Other: Crisis Response Planning intervention (structures safety planning) — Collaborative safety planning intervention delivered by trained clinical psychologists in 20-45 minute sessions. Participants create personalized, written crisis response plans identifying warning signs of emotional distress, internal coping strategies, social support contacts, professional resources, and means restriction methods. The intervention follows a structured format focusing on practical crisis management tools that participants can implement during suicidal crises.
  Arms: Crisis Response Planning plus Optimized Usual Treatment; Optimized Usual Treatment Only

SUMMARY:
1. Background Suicide is a major public health challenge with over 800,000 deaths annually worldwide. Brazil experienced a concerning 57% increase in suicide rates between 2000-2019, highlighting urgent need for effective prevention strategies. This study evaluates two promising interventions: esketamine (rapid-acting pharmacological treatment) and Crisis Response Planning (CRP, evidence-based psychological safety planning approach) in a real-world Brazilian public health setting.
2. Study Design

   Pragmatic randomized controlled trial with hybrid implementation-effectiveness design comparing three approaches in emergency departments across two Brazilian cities with combined population of 310,000:
   * Group A: Single esketamine infusion (0.5 mg/kg over 40 minutes) + optimized usual treatment (OUT)
   * Group B: Crisis Response Planning + OUT
   * Group C: OUT alone (enhanced control)
3. Participants

   Adults and adolescents (≥14 years) presenting with high suicide risk defined as:
   * Recent suicide attempts within 30 days (actual, interrupted, or aborted)
   * Severe suicidal ideation (Columbia-Suicide Severity Rating Scale questions 4-5 positive)
   * Non-suicidal self-harm requiring emergency medical attention
4. Target enrollment: ~272 participants per group (816 total). Key exclusions: esketamine contraindications (cardiovascular disease, aneurysms), psychotic disorders, severe substance use disorders, pregnancy/lactation, inability to consent.
5. Interventions

   1. Esketamine Group: IV infusion administered in medical setting with continuous 4-hour monitoring (pulse, blood pressure, ECG, oxygen saturation). Trained medical staff and emergency protocols available.
   2. Crisis Response Planning: Collaborative intervention delivered by trained clinical psychologists. 20-45 minute sessions creating personalized, written safety plans identifying warning signs, internal coping strategies, social support contacts, professional resources, and means restriction.
   3. Optimized Usual Treatment: Enhanced standard care including guaranteed psychiatric follow-up appointment within one week through municipal mental health services (CAPS - Psychosocial Care Centers).
6. Primary Outcome Repeated suicide-related events over one year including suicide attempts, interrupted attempts, suicide-prevention hospitalizations, deaths by suicide, and non-suicidal self-harm requiring medical attention.
7. Comprehensive Data Collection

   1. Biomarkers: 10mL venous blood samples (2 EDTA tubes) collected at baseline by senior clinical nurses. Comprehensive laboratory analysis including complete blood count, metabolic panel, vitamins (B1, B2, B6, B12, B9, D, K), hormones (TSH, T3, T4, testosterone, DHEA, prolactin), inflammatory markers (CRP), brain-derived neurotrophic factor (BDNF), platelet monoamine oxidase (MAO), minerals (iron, ferritin, magnesium, zinc, selenium), and lipid profiles. Samples processed within 24 hours and stored at -80°C for analysis.
   2. Clinical Assessments: Comprehensive evaluations at 11 time points (baseline, 24 hours, 7 days, 2 weeks, 4 weeks, 8 weeks, 16 weeks, 24 weeks, 32 weeks, 40 weeks, 1 year) using validated instruments: Columbia-Suicide Severity Rating Scale (C-SSRS), depression scales (PHQ-9, MADRS), anxiety (GAD-7), quality of life (SF-36v2), impulsivity (BIS-11), trauma history (MACE), substance use (ASSIST), sleep quality (PSQI), and additional psychosocial measures.
   3. Ecological Momentary Assessment: Real-time data collection via smartphone application for consenting participants. Six daily prompts assessing mood, suicidal thoughts, and emotional states using validated scales. Previous research demonstrates safety and high compliance rates in suicide research populations.
8. Secondary Outcomes

   * Time to new suicidal crisis or psychiatric emergency
   * Changes in depression and anxiety severity scores
   * Quality of life and functional outcome improvements
   * Treatment response variability by demographic factors (age, gender, socioeconomic status)
   * Comprehensive cost-effectiveness analysis including direct medical costs and indirect productivity losses
   * Patient and clinician satisfaction with treatment modalities
   * Implementation barriers and facilitators using Consolidated Framework for Implementation Research (CFIR)
   * Biomarker predictors of treatment response
9. Clinical Significance This represents the first large-scale, real-world direct comparison of rapid-acting pharmacological (esketamine) versus evidence-based psychological (CRP) interventions for suicide prevention within a public health system. Results will provide crucial evidence for clinical practice guidelines and inform implementation of these interventions in Brazil and similar global contexts. The pragmatic design ensures findings are directly applicable to routine emergency department practice, while comprehensive biomarker analysis may identify biological predictors of treatment response to personalize suicide prevention approaches.

DETAILED DESCRIPTION:
Additional Open-Label Study for Recurrent Suicide: Any participant who experiences a recurrent suicidal crisis-thus meeting the primary outcome of the study-will be eligible to participate in a secondary open-label study (ketamine + CRP + OUT). In this phase, participants will be treated and followed for the remainder of the 1-year period.

ELIGIBILITY:
* Inclusion Criteria:

  * Age ≥ 14 years
  * Recent suicide attempt within 30 days (actual, interrupted, or aborted)
  * Severe suicidal ideation (positive response to questions 4 or 5 on Columbia-Suicide Severity Rating Scale screening version)
  * Non-suicidal self-harm requiring medical attention in emergency department setting
  * Resident of Jaguariúna, Indaiatuba, or surrounding areas
  * Able to provide informed consent (or assent with guardian consent for minors)
  * Not requiring long-term psychiatric hospitalization after emergency evaluation
* Exclusion Criteria:

  * Medical conditions contraindicated for esketamine use (aneurysmal vascular disease, arteriovenous malformation, intracerebral hemorrhage, known hypersensitivity to esketamine)
  * Need for intensive care unit admission without possibility of later study participation
  * Severe substance use disorders interfering with protocol adherence
  * Psychotic disorders
  * Lack of stable housing or inability to be contacted for follow-up assessments
  * History of non-response to esketamine or previous enrollment in esketamine studies
  * Pregnancy or breastfeeding
  * Inability to provide informed consent due to cognitive impairment or explicit refusal to participate

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Repeated Suicide-Related Events at One Year | One year from baseline enrollment
  Composite outcome including repeated suicide attempts (actual, interrupted, aborted), hospitalizations for suicide prevention, deaths by suicide, and non-suicidal self-harm requiring medical attention in emergency settings. Based on validated definitions from the Columbia-Suicide Severity Rating Scale and previous suicide prevention studies. Events assessed through medical records review, participant self-report, and contact with emergency services in both study municipalities.

SECONDARY OUTCOMES:
Changes in Depressive Symptoms and Depression Prevalence | Baseline, 7 days, 1 month, 3 months, 6 months, and 1 year
  Changes in mental health scores measured by Patient Health Questionnaire-9 (PHQ-9), assessed at multiple time points to evaluate treatment impact on overall mental health status.
Changes in Depressive Symptoms and Depression Prevalence | Baseline, 7 days, 1 month, 3 months, 6 months, and 1 year
  Changes in mental health scores measured by Montgomery-Asberg Depression Rating Scale (MADRS), assessed at multiple time points to evaluate treatment impact on overall mental health status.
Changes in Depression, Anxiety, and Mood Disorder Severity | Baseline, 7 days, 1 month, 3 months, 6 months, and 1 year
  Changes in mental health scores measured by Generalized Anxiety Disorder-7 (GAD-7), assessed at multiple time points to evaluate treatment impact on overall mental health status.
Changes in Depression, Anxiety, and Mood Disorder Severity | Baseline, 7 days, 1 month, 3 months, 6 months, and 1 year
  Changes in mental health scores measured by the Hypomania Checklist (HCL-32) Questionnaire, assessed at multiple time points to evaluate treatment impact on overall mental health status.
Time to Next Suicidal Crisis or Emergency | Up to one year from baseline
  Time elapsed between initial intervention and occurrence of any new suicidal crisis, including suicide attempts, hospitalization, or emergency department visits related to suicidal behavior. Measured using survival analysis methods with censoring at study completion.
Demographic Variability in Treatment Response | One year from baseline
  Analysis of treatment outcome differences across demographic subgroups including age, gender, socioeconomic status, and other baseline characteristics. Identifies which populations may benefit most from specific interventions.
Changes in Patient-Reported Quality of Life | Baseline, 1 month, 3 months, 6 months, and 1 year
  Changes in quality of life measured by SF-36v2 questionnaire, assessed at multiple timepoints.
Frequency and Nature of Treatment-Related Adverse Events | Throughout study participation, up to one year
  Documentation of all adverse events, complications, and safety concerns associated with each treatment arm, including physical symptoms after esketamine infusion, psychological distress during crisis planning sessions, and any serious adverse events.
Comparative Cost-Effectiveness of Treatment Approaches | One year from baseline enrollment
  Economic evaluation comparing direct medical costs, indirect productivity losses, healthcare utilization, and cost per quality-adjusted life year (QALY) across treatment groups. Includes medication costs, therapy sessions, hospitalizations, and lost productivity.
Patients' Treatment Satisfaction and Acceptability Ratings | 1 month, 6 months, and 1 year post-treatment
  Patients' satisfaction scores evaluating perceived effectiveness, feasibility, and acceptability of each treatment modality, assessed through qualitative interviews.
Healthcare Providers' Treatment Satisfaction and Acceptability Ratings | 1 month, 6 months, and 1 year post-treatment
  Healthcare Providers' satisfaction scores evaluating perceived effectiveness, feasibility, and acceptability of each treatment modality, assessed through qualitative interviews.
Implementation Science Outcomes for Clinical Integration | Throughout study conduct, analyzed at study completion
  Identification of barriers and facilitators for implementing esketamine therapy and crisis response planning in emergency department settings, evaluated using the Consolidated Framework for Implementation Research (CFIR).
Post-Treatment Healthcare Service Utilization | Six months and one year post-treatment
  Comparison of readmission rates, additional mental health service needs, emergency department visits, and psychiatric consultations across treatment groups during follow-up period.
Healthcare Professional Engagement with Implementation Strategies | Throughout study conduct, up to one year
  Rate of healthcare professional adherence to implementation strategies, engagement with training programs, and adoption of study interventions in routine clinical practice within the emergency department settings.
Serum Brain-derived neurotrophic factor (BDNF) Predictor of Treatment Outcome | Baseline biomarker collection with outcome correlation at 6 months and 1 year
  Analysis of baseline serum Brain-derived neurotrophic factor (BDNF) as a predictor of treatment response and resistance. Identifies biological factors that may guide personalized treatment selection.
Monoamine oxidase (MAO) Predictor of Treatment Outcome | Baseline biomarker collection with outcome correlation at 6 months and 1 year
  Analysis of baseline platelet Monoamine oxidase (MAO) as a predictor of treatment response and resistance. Identifies biological factors that may guide personalized treatment selection.
Hormones (TSH, T3, Free T3 and Free T4, Total Testosterone, SHBG, S-DHEA, Prolactin) Predictors of Treatment Outcome | Baseline biomarker collection with outcome correlation at 6 months and 1 year
  Analysis of baseline hormones (TSH, T3, Free T3 and Free T4, Total Testosterone, SHBG, S-DHEA, Prolactin) as predictors of treatment response and resistance. Identifies biological factors that may guide personalized treatment selection.
Vitamins and Minerals Biomarkers Predictors of Treatment Outcome | Baseline biomarker collection with outcome correlation at 6 months and 1 year
  Analysis of baseline vitamins and minerals (25-hydroxy-vitamin D, Vitamin B1, Vitamin B12, Vitamin B6, and Folic Acid (B9), Vitamin K, Magnesium, and Red Blood Cell/Erythrocyte Zinc) as predictors of treatment response and resistance. Identifies biological factors that may guide personalized treatment selection.
Iron Profile (Iron, Ferritin and Transferrin Saturation) Predictors of Treatment Outcome | Baseline biomarker collection with outcome correlation at 6 months and 1 year
  Analysis of baseline Iron Profile (Iron, Ferritin, and Transferrin Saturation) as predictors of treatment response and resistance. Identifies biological factors that may guide personalized treatment selection.
Homocysteine Predictor of Treatment Outcome | Baseline biomarker collection with outcome correlation at 6 months and 1 year
  Analysis of baseline Homocysteine as a predictor of treatment response and resistance. Identifies biological factors that may guide personalized treatment selection.
Ultrasensitive C-Reactive Protein Predictor of Treatment Outcome | Baseline biomarker collection with outcome correlation at 6 months and 1 year
  Analysis of baseline Ultrasensitive C-Reactive Protein as a predictor of treatment response and resistance. Identifies biological factors that may guide personalized treatment selection.
25-hydroxy-vitamin D Predictor of Treatment Outcome | Baseline biomarker collection with outcome correlation at 6 months and 1 year
  Analysis of baseline 25-hydroxy-vitamin D as a predictor of treatment response and resistance. Identifies biological factors that may guide personalized treatment selection.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and confidentiality, particularly given the sensitive nature of suicide-related data and the vulnerable population being studied. The study involves detailed mental health assessments, suicide risk evaluations, and personal crisis information that requires strict confidentiality protections under Brazilian data protection laws and research ethics guidelines.
  Aggregate, de-identified results and statistical analyses will be made available through peer-reviewed publications and conference presentations. Researchers interested in collaboration or secondary analyses may contact the principal investigator to discuss potential partnerships within appropriate ethical and regulatory frameworks.
  The study protocol, statistical analysis plan, and aggregate results will be made publicly available to support scientific transparency while maintaining participant confidentiality.

REFERENCES:
- [Background] Zisook S, Domingues I, Compton J. Pharmacologic Approaches to Suicide Prevention. Focus (Am Psychiatr Publ). 2023 Apr;21(2):137-144. doi: 10.1176/appi.focus.20220076. Epub 2023 Apr 14. PMID 37201142
- [Background] Zimmerman M, Balling C. Screening for Borderline Personality Disorder With the McLean Screening Instrument: A Review and Critique of the Literature. J Pers Disord. 2021 Apr;35(2):288-298. doi: 10.1521/pedi_2019_33_451. Epub 2019 Dec 30. PMID 31887102
- [Background] Zanos P, Gould TD. Mechanisms of ketamine action as an antidepressant. Mol Psychiatry. 2018 Apr;23(4):801-811. doi: 10.1038/mp.2017.255. Epub 2018 Mar 13. PMID 29532791
- [Background] Zalsman G, Hawton K, Wasserman D, van Heeringen K, Arensman E, Sarchiapone M, Carli V, Hoschl C, Barzilay R, Balazs J, Purebl G, Kahn JP, Saiz PA, Lipsicas CB, Bobes J, Cozman D, Hegerl U, Zohar J. Suicide prevention strategies revisited: 10-year systematic review. Lancet Psychiatry. 2016 Jul;3(7):646-59. doi: 10.1016/S2215-0366(16)30030-X. Epub 2016 Jun 8. PMID 27289303
- [Background] Zaki N, Chen LN, Lane R, Doherty T, Drevets WC, Morrison RL, Sanacora G, Wilkinson ST, Popova V, Fu DJ. Long-term safety and maintenance of response with esketamine nasal spray in participants with treatment-resistant depression: interim results of the SUSTAIN-3 study. Neuropsychopharmacology. 2023 Jul;48(8):1225-1233. doi: 10.1038/s41386-023-01577-5. Epub 2023 May 12. PMID 37173512
- [Background] Wu H, Lu L, Qian Y, Jin XH, Yu HR, Du L, Fu XL, Zhu B, Chen HL. The significance of cognitive-behavioral therapy on suicide: An umbrella review. J Affect Disord. 2022 Nov 15;317:142-148. doi: 10.1016/j.jad.2022.08.067. Epub 2022 Aug 27. PMID 36041581
- [Background] Wittkampf KA, Naeije L, Schene AH, Huyser J, van Weert HC. Diagnostic accuracy of the mood module of the Patient Health Questionnaire: a systematic review. Gen Hosp Psychiatry. 2007 Sep-Oct;29(5):388-95. doi: 10.1016/j.genhosppsych.2007.06.004. PMID 17888804
- [Background] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Background] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Pharmacological interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Jan 10;1(1):CD013669. doi: 10.1002/14651858.CD013669.pub2. PMID 35608866
- [Background] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Background] Witt A, Ordonez A, Martin A, Vitiello B, Fegert JM. Child and adolescent mental health service provision and research during the Covid-19 pandemic: challenges, opportunities, and a call for submissions. Child Adolesc Psychiatry Ment Health. 2020 May 11;14:19. doi: 10.1186/s13034-020-00324-8. eCollection 2020. No abstract available. PMID 32411296
- [Background] Wilkinson ST, Trujillo Diaz D, Rupp ZW, Kidambi A, Ramirez KL, Flores JM, Avila-Quintero VJ, Rhee TG, Olfson M, Bloch MH. Pharmacological and somatic treatment effects on suicide in adults: A systematic review and meta-analysis. Depress Anxiety. 2022 Feb;39(2):100-112. doi: 10.1002/da.23222. Epub 2021 Nov 11. PMID 34762330
- [Background] Wilkinson ST, Ballard ED, Bloch MH, Mathew SJ, Murrough JW, Feder A, Sos P, Wang G, Zarate CA Jr, Sanacora G. The Effect of a Single Dose of Intravenous Ketamine on Suicidal Ideation: A Systematic Review and Individual Participant Data Meta-Analysis. Am J Psychiatry. 2018 Feb 1;175(2):150-158. doi: 10.1176/appi.ajp.2017.17040472. Epub 2017 Oct 3. PMID 28969441
- [Background] WHO (2016). Global Health Observatory (GHO) Data: Suicide Rates. Geneva, Switzerland, World Health Organization
- [Background] WHO (2014). Preventing suicide: A global imperative: 92.
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Ward-Ciesielski EF, Schumacher JA, Bagge CL. Relations Between Nonsuicidal Self-Injury and Suicide Attempt Characteristics in a Sample of Recent Suicide Attempters. Crisis. 2016 Jul;37(4):310-313. doi: 10.1027/0227-5910/a000400. Epub 2016 Jun 24. PMID 27338291
- [Background] Wang C, Zhou Y, Zheng W, Liu W, Zhan Y, Li H, Chen L, Zhang B, Walter M, Li M, Li MD, Ning Y. Association between depression subtypes and response to repeated-dose intravenous ketamine. Acta Psychiatr Scand. 2019 Nov;140(5):446-457. doi: 10.1111/acps.13096. Epub 2019 Sep 20. PMID 31483855
- [Background] Wagner E, Kane JM, Correll CU, Howes O, Siskind D, Honer WG, Lee J, Falkai P, Schneider-Axmann T, Hasan A; TRRIP Working Group. Clozapine Combination and Augmentation Strategies in Patients With Schizophrenia -Recommendations From an International Expert Survey Among the Treatment Response and Resistance in Psychosis (TRRIP) Working Group. Schizophr Bull. 2020 Dec 1;46(6):1459-1470. doi: 10.1093/schbul/sbaa060. PMID 32421188
- [Background] Victor SE, Klonsky ED. Correlates of suicide attempts among self-injurers: a meta-analysis. Clin Psychol Rev. 2014 Jun;34(4):282-97. doi: 10.1016/j.cpr.2014.03.005. Epub 2014 Apr 2. PMID 24742496
- [Background] Vermeulen JM, van Rooijen G, van de Kerkhof MPJ, Sutterland AL, Correll CU, de Haan L. Clozapine and Long-Term Mortality Risk in Patients With Schizophrenia: A Systematic Review and Meta-analysis of Studies Lasting 1.1-12.5 Years. Schizophr Bull. 2019 Mar 7;45(2):315-329. doi: 10.1093/schbul/sby052. PMID 29697804
- [Background] Turkoz I, Nelson JC, Wilkinson ST, Borentain S, Macaluso M, Trivedi MH, Williamson D, Sheehan JJ, Salvadore G, Singh J, Daly E. Predictors of response and remission in patients with treatment-resistant depression: A post hoc pooled analysis of two acute trials of esketamine nasal spray. Psychiatry Res. 2023 May;323:115165. doi: 10.1016/j.psychres.2023.115165. Epub 2023 Mar 16. PMID 37019044
- [Background] Trull TJ, Ebner-Priemer UW. Using experience sampling methods/ecological momentary assessment (ESM/EMA) in clinical assessment and clinical research: introduction to the special section. Psychol Assess. 2009 Dec;21(4):457-62. doi: 10.1037/a0017653. PMID 19947780
- [Background] Taylor GJ, Ryan D, Bagby RM. Toward the development of a new self-report alexithymia scale. Psychother Psychosom. 1985;44(4):191-9. doi: 10.1159/000287912. PMID 3837277
- [Background] Sufrate-Sorzano T, Santolalla-Arnedo I, Garrote-Camara ME, Angulo-Nalda B, Cotelo-Saenz R, Pastells-Peiro R, Bellon F, Blanco-Blanco J, Juarez-Vela R, Molina-Luque F. Interventions of choice for the prevention and treatment of suicidal behaviours: An umbrella review. Nurs Open. 2023 Aug;10(8):4959-4970. doi: 10.1002/nop2.1820. Epub 2023 May 22. PMID 37218123
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Stanley B, Brown GK, Brenner LA, Galfalvy HC, Currier GW, Knox KL, Chaudhury SR, Bush AL, Green KL. Comparison of the Safety Planning Intervention With Follow-up vs Usual Care of Suicidal Patients Treated in the Emergency Department. JAMA Psychiatry. 2018 Sep 1;75(9):894-900. doi: 10.1001/jamapsychiatry.2018.1776. PMID 29998307
- [Background] Stanley, B. and G. K. Brown (2012). "Safety Planning Intervention: A Brief Intervention to Mitigate Suicide Risk." Cognitive and Behavioral Practice 19(2): 256-264
- [Background] Spitzer RL, Williams JB, Kroenke K, Linzer M, deGruy FV 3rd, Hahn SR, Brody D, Johnson JG. Utility of a new procedure for diagnosing mental disorders in primary care. The PRIME-MD 1000 study. JAMA. 1994 Dec 14;272(22):1749-56. PMID 7966923
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Smith KA, Cipriani A. Lithium and suicide in mood disorders: Updated meta-review of the scientific literature. Bipolar Disord. 2017 Nov;19(7):575-586. doi: 10.1111/bdi.12543. Epub 2017 Sep 12. PMID 28895269
- [Background] Siegel AN, Di Vincenzo JD, Brietzke E, Gill H, Rodrigues NB, Lui LMW, Teopiz KM, Ng J, Ho R, McIntyre RS, Rosenblat JD. Antisuicidal and antidepressant effects of ketamine and esketamine in patients with baseline suicidality: A systematic review. J Psychiatr Res. 2021 May;137:426-436. doi: 10.1016/j.jpsychires.2021.03.009. Epub 2021 Mar 16. PMID 33774537
- [Background] Short B, Fong J, Galvez V, Shelker W, Loo CK. Side-effects associated with ketamine use in depression: a systematic review. Lancet Psychiatry. 2018 Jan;5(1):65-78. doi: 10.1016/S2215-0366(17)30272-9. Epub 2017 Jul 27. PMID 28757132
- [Background] Shivanekar S, Gopalan P, Pizon A, Spotts C, Cruz N, Lightfoot M, Rohac R, Baumeister A, Griffo A, Panny B, Kucherer S, Israel A, Rengasamy M, Price R. A Pilot Study of Ketamine Infusion after Suicide Attempt: New Frontiers in Treating Acute Suicidality in a Real-World Medical Setting. Int J Environ Res Public Health. 2022 Oct 24;19(21):13792. doi: 10.3390/ijerph192113792. PMID 36360672
- [Background] Shepard DS, Gurewich D, Lwin AK, Reed GA Jr, Silverman MM. Suicide and Suicidal Attempts in the United States: Costs and Policy Implications. Suicide Life Threat Behav. 2016 Jun;46(3):352-62. doi: 10.1111/sltb.12225. Epub 2015 Oct 29. PMID 26511788
- [Background] Shen Z, Gao D, Lv X, Wang H, Yue W. A meta-analysis of the effects of ketamine on suicidal ideation in depression patients. Transl Psychiatry. 2024 Jun 10;14(1):248. doi: 10.1038/s41398-024-02973-1. PMID 38858391
- [Background] Sgobin SM, Traballi AL, Botega NJ, Coelho OR. Direct and indirect cost of attempted suicide in a general hospital: cost-of-illness study. Sao Paulo Med J. 2015 May-Jun;133(3):218-26. doi: 10.1590/1516-3180.2014.8491808. Epub 2015 Jun 1. PMID 26176926
- [Background] Santos JJ, Costa TA, Guilherme JH, Silva WC, Abentroth LR, Krebs JA, Sotoriva P. Adaptation and cross-cultural validation of the Brazilian version of the Warwick-Edinburgh mental well-being scale. Rev Assoc Med Bras (1992). 2015 May-Jun;61(3):209-14. doi: 10.1590/1806-9282.61.03.209. PMID 26248241
- [Background] Rudd MD, Mandrusiak M, Joiner TE Jr. The case against no-suicide contracts: the commitment to treatment statement as a practice alternative. J Clin Psychol. 2006 Feb;62(2):243-51. doi: 10.1002/jclp.20227. PMID 16342293
- [Background] Rozek DC, Keane C, Sippel LM, Stein JY, Rollo-Carlson C, Bryan CJ. Short-term effects of crisis response planning on optimism in a U.S. Army sample. Early Interv Psychiatry. 2019 Jun;13(3):682-685. doi: 10.1111/eip.12699. Epub 2018 Jun 26. PMID 29943518
- [Background] Rozek DC, Bryan CJ. Integrating crisis response planning for suicide prevention into trauma-focused treatments: A military case example. J Clin Psychol. 2020 May;76(5):852-864. doi: 10.1002/jclp.22920. Epub 2020 Jan 11. PMID 31926024
- [Background] Rong C, Park C, Rosenblat JD, Subramaniapillai M, Zuckerman H, Fus D, Lee YL, Pan Z, Brietzke E, Mansur RB, Cha DS, Lui LMW, McIntyre RS. Predictors of Response to Ketamine in Treatment Resistant Major Depressive Disorder and Bipolar Disorder. Int J Environ Res Public Health. 2018 Apr 17;15(4):771. doi: 10.3390/ijerph15040771. PMID 29673146
- [Background] Quinlivan L, Cooper J, Davies L, Hawton K, Gunnell D, Kapur N. Which are the most useful scales for predicting repeat self-harm? A systematic review evaluating risk scales using measures of diagnostic accuracy. BMJ Open. 2016 Feb 12;6(2):e009297. doi: 10.1136/bmjopen-2015-009297. PMID 26873046
- [Background] Pretorius TB, Padmanabhanunni A. A unidimensional short form of the Beck Hopelessness Scale (BHS-7) derived using item response theory. Sci Rep. 2024 Mar 12;14(1):6021. doi: 10.1038/s41598-024-56792-x. PMID 38472416
- [Background] Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry. 2007 Jul;164(7):1035-43. doi: 10.1176/ajp.2007.164.7.1035. PMID 17606655
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124
- [Background] Park LT, Luckenbaugh DA, Pennybaker SJ, Hopkins MA, Henter ID, Lener MS, Kadriu B, Ballard ED, Zarate CA Jr. The effects of ketamine on typical and atypical depressive symptoms. Acta Psychiatr Scand. 2020 Nov;142(5):394-401. doi: 10.1111/acps.13216. Epub 2020 Aug 6. PMID 32677051
- [Background] Pan Y, Gorenflo MP, Davis PB, Kaelber DC, De Luca S, Xu R. Suicidal ideation following ketamine prescription in patients with recurrent major depressive disorder: a nation-wide cohort study. Transl Psychiatry. 2024 Aug 9;14(1):327. doi: 10.1038/s41398-024-03033-4. PMID 39122686
- [Background] Oquendo MA, Galfalvy HC, Choo TH, Herzog S, Burke AK, Sublette ME, Mann JJ, Stanley BH. Occurrence and characteristics of suicidal ideation in psychiatrically healthy individuals based on ecological momentary assessment. Mol Psychiatry. 2024 Nov;29(11):3356-3363. doi: 10.1038/s41380-024-02560-2. Epub 2024 May 10. PMID 38729992
- [Background] Nock MK, Holmberg EB, Photos VI, Michel BD. Self-Injurious Thoughts and Behaviors Interview: development, reliability, and validity in an adolescent sample. Psychol Assess. 2007 Sep;19(3):309-17. doi: 10.1037/1040-3590.19.3.309. PMID 17845122
- [Background] Nikayin S, Murphy E, Krystal JH, Wilkinson ST. Long-term safety of ketamine and esketamine in treatment of depression. Expert Opin Drug Saf. 2022 Jun;21(6):777-787. doi: 10.1080/14740338.2022.2066651. Epub 2022 Apr 19. PMID 35416105
- [Background] Ngin NLX, Hassan NB, Koh SLS. Predicting suicide and suicide attempts in adults in acute hospitals: A systematic review of diagnostic accuracy evaluating risk scales. Int J Nurs Stud. 2022 Dec;136:104361. doi: 10.1016/j.ijnurstu.2022.104361. Epub 2022 Sep 16. PMID 36209575
- [Background] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Background] Mendez-Bustos P, Calati R, Rubio-Ramirez F, Olie E, Courtet P, Lopez-Castroman J. Effectiveness of Psychotherapy on Suicidal Risk: A Systematic Review of Observational Studies. Front Psychol. 2019 Feb 19;10:277. doi: 10.3389/fpsyg.2019.00277. eCollection 2019. PMID 30837920
- [Background] Medeiros GC, Gould TD, Prueitt WL, Nanavati J, Grunebaum MF, Farber NB, Singh B, Selvaraj S, Machado-Vieira R, Achtyes ED, Parikh SV, Frye MA, Zarate CA Jr, Goes FS. Blood-based biomarkers of antidepressant response to ketamine and esketamine: A systematic review and meta-analysis. Mol Psychiatry. 2022 Sep;27(9):3658-3669. doi: 10.1038/s41380-022-01652-1. Epub 2022 Jun 27. PMID 35760879
- [Background] McInnes LA, Qian JJ, Gargeya RS, DeBattista C, Heifets BD. A retrospective analysis of ketamine intravenous therapy for depression in real-world care settings. J Affect Disord. 2022 Mar 15;301:486-495. doi: 10.1016/j.jad.2021.12.097. Epub 2022 Jan 11. PMID 35027209
- [Background] Zanarini MC, Vujanovic AA, Parachini EA, Boulanger JL, Frankenburg FR, Hennen J. A screening measure for BPD: the McLean Screening Instrument for Borderline Personality Disorder (MSI-BPD). J Pers Disord. 2003 Dec;17(6):568-73. doi: 10.1521/pedi.17.6.568.25355. PMID 14744082
- [Background] Mann JJ, Michel CA, Auerbach RP. Improving Suicide Prevention Through Evidence-Based Strategies: A Systematic Review. Am J Psychiatry. 2021 Jul;178(7):611-624. doi: 10.1176/appi.ajp.2020.20060864. Epub 2021 Feb 18. PMID 33596680
- [Background] Mancuso E, Sampogna G, Boiano A, Della Rocca B, Di Vincenzo M, Lapadula MV, Martinelli F, Lucci F, Luciano M. Biological correlates of treatment resistant depression: a review of peripheral biomarkers. Front Psychiatry. 2023 Oct 24;14:1291176. doi: 10.3389/fpsyt.2023.1291176. eCollection 2023. PMID 37941970
- [Background] Mamdani F, Weber MD, Bunney B, Burke K, Cartagena P, Walsh D, Lee FS, Barchas J, Schatzberg AF, Myers RM, Watson SJ, Akil H, Vawter MP, Bunney WE, Sequeira A. Identification of potential blood biomarkers associated with suicide in major depressive disorder. Transl Psychiatry. 2022 Apr 14;12(1):159. doi: 10.1038/s41398-022-01918-w. PMID 35422091
- [Background] Malloy-Diniz LF, Paula JJ, Vasconcelos AG, Almondes KM, Pessoa R, Faria L, Coutinho G, Costa DS, Duran V, Coutinho TV, Correa H, Fuentes D, Abreu N, Mattos P. Normative data of the Barratt Impulsiveness Scale 11 (BIS-11) for Brazilian adults. Braz J Psychiatry. 2015 Jul-Sep;37(3):245-8. doi: 10.1590/1516-4446-2014-1599. PMID 26376056
- [Background] Malloy-Diniz, L. F., P. Mattos, W. B. Leite, N. Abreu, G. Coutinho, J. J. d. Paula, H. Tavares, A. G. Vasconcelos and D. Fuentes (2010). "Tradução e adaptação cultural da Barratt Impulsiveness Scale (BIS-11) para aplicação em adultos brasileiros." Jornal Brasileiro de Psiquiatria 59: 99-105
- [Background] Lucchetti G, Granero Lucchetti AL, Peres MF, Leao FC, Moreira-Almeida A, Koenig HG. Validation of the Duke Religion Index: DUREL (Portuguese version). J Relig Health. 2012 Jun;51(2):579-86. doi: 10.1007/s10943-010-9429-5. PMID 21107911
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Krystal JH, Kavalali ET, Monteggia LM. Ketamine and rapid antidepressant action: new treatments and novel synaptic signaling mechanisms. Neuropsychopharmacology. 2024 Jan;49(1):41-50. doi: 10.1038/s41386-023-01629-w. Epub 2023 Jul 24. PMID 37488280
- [Background] Koenig H, Parkerson GR Jr, Meador KG. Religion index for psychiatric research. Am J Psychiatry. 1997 Jun;154(6):885-6. doi: 10.1176/ajp.154.6.885b. No abstract available. PMID 9167530
- [Background] Klonsky ED, Glenn CR. Assessing the functions of non-suicidal self-injury: Psychometric properties of the Inventory of Statements About Self-injury (ISAS). J Psychopathol Behav Assess. 2009 Sep;31(3):215-219. doi: 10.1007/s10862-008-9107-z. Epub 2008 Oct 30. PMID 29269992
- [Background] Kivela L, van der Does WAJ, Riese H, Antypa N. Don't Miss the Moment: A Systematic Review of Ecological Momentary Assessment in Suicide Research. Front Digit Health. 2022 May 6;4:876595. doi: 10.3389/fdgth.2022.876595. eCollection 2022. PMID 35601888
- [Background] Katz IR, Rogers MP, Lew R, Thwin SS, Doros G, Ahearn E, Ostacher MJ, DeLisi LE, Smith EG, Ringer RJ, Ferguson R, Hoffman B, Kaufman JS, Paik JM, Conrad CH, Holmberg EF, Boney TY, Huang GD, Liang MH; Li+ plus Investigators. Lithium Treatment in the Prevention of Repeat Suicide-Related Outcomes in Veterans With Major Depression or Bipolar Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Jan 1;79(1):24-32. doi: 10.1001/jamapsychiatry.2021.3170. PMID 34787653
- [Background] Johnston JN, Campbell D, Caruncho HJ, Henter ID, Ballard ED, Zarate CA. Suicide Biomarkers to Predict Risk, Classify Diagnostic Subtypes, and Identify Novel Therapeutic Targets: 5 Years of Promising Research. Int J Neuropsychopharmacol. 2022 Mar 17;25(3):197-214. doi: 10.1093/ijnp/pyab083. PMID 34865007
- [Background] Jesus-Nunes AP, Leal GC, Correia-Melo FS, Vieira F, Mello RP, Caliman-Fontes AT, Echegaray MVF, Marback RF, Guerreiro-Costa LNF, Souza-Marques B, Santos-Lima C, Souza LS, Bandeira ID, Kapczinski F, Lacerda ALT, Quarantini LC. Clinical predictors of depressive symptom remission and response after racemic ketamine and esketamine infusion in treatment-resistant depression. Hum Psychopharmacol. 2022 Jul;37(4):e2836. doi: 10.1002/hup.2836. Epub 2022 Feb 18. PMID 35179810
- [Background] Inagaki M, Kawashima Y, Yonemoto N, Yamada M. Active contact and follow-up interventions to prevent repeat suicide attempts during high-risk periods among patients admitted to emergency departments for suicidal behavior: a systematic review and meta-analysis. BMC Psychiatry. 2019 Jan 25;19(1):44. doi: 10.1186/s12888-019-2017-7. PMID 30683075
- [Background] Inagaki M, Kawashima Y, Kawanishi C, Yonemoto N, Sugimoto T, Furuno T, Ikeshita K, Eto N, Tachikawa H, Shiraishi Y, Yamada M. Interventions to prevent repeat suicidal behavior in patients admitted to an emergency department for a suicide attempt: a meta-analysis. J Affect Disord. 2015 Apr 1;175:66-78. doi: 10.1016/j.jad.2014.12.048. Epub 2014 Dec 30. PMID 25594513
- [Background] Humeniuk R, Ali R, Babor TF, Farrell M, Formigoni ML, Jittiwutikarn J, de Lacerda RB, Ling W, Marsden J, Monteiro M, Nhiwatiwa S, Pal H, Poznyak V, Simon S. Validation of the Alcohol, Smoking And Substance Involvement Screening Test (ASSIST). Addiction. 2008 Jun;103(6):1039-47. doi: 10.1111/j.1360-0443.2007.02114.x. Epub 2008 Mar 28. PMID 18373724
- [Background] Hochschild A, Grunebaum MF, Mann JJ. The rapid anti-suicidal ideation effect of ketamine: A systematic review. Prev Med. 2021 Nov;152(Pt 1):106524. doi: 10.1016/j.ypmed.2021.106524. Epub 2021 Sep 16. PMID 34538369
- [Background] Hietamies TM, McInnes LA, Klise AJ, Worley MJ, Qian JJ, Williams LM, Heifets BD, Levine SP. The effects of ketamine on symptoms of depression and anxiety in real-world care settings: A retrospective controlled analysis. J Affect Disord. 2023 Aug 15;335:484-492. doi: 10.1016/j.jad.2023.04.141. Epub 2023 May 16. PMID 37201900
- [Background] Henrique IF, De Micheli D, Lacerda RB, Lacerda LA, Formigoni ML. [Validation of the Brazilian version of Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)]. Rev Assoc Med Bras (1992). 2004 Apr-Jun;50(2):199-206. doi: 10.1590/s0104-42302004000200039. Epub 2004 Jul 21. Portuguese. PMID 15286871
- [Background] Harris IM, Beese S, Moore D. Predicting repeated self-harm or suicide in adolescents and young adults using risk assessment scales/tools: a systematic review protocol. Syst Rev. 2019 Apr 4;8(1):87. doi: 10.1186/s13643-019-1007-7. PMID 30947743
- [Background] Harris IM, Beese S, Moore D. Predicting future self-harm or suicide in adolescents: a systematic review of risk assessment scales/tools. BMJ Open. 2019 Sep 6;9(9):e029311. doi: 10.1136/bmjopen-2019-029311. PMID 31494608
- [Background] Haile CN, Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Foulkes A, Iqbal S, Mahoney JJ 3rd, De La Garza R 2nd, Charney DS, Newton TF, Mathew SJ. Plasma brain derived neurotrophic factor (BDNF) and response to ketamine in treatment-resistant depression. Int J Neuropsychopharmacol. 2014 Feb;17(2):331-6. doi: 10.1017/S1461145713001119. Epub 2013 Oct 8. PMID 24103211
- [Background] WHO ASSIST Working Group. The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): development, reliability and feasibility. Addiction. 2002 Sep;97(9):1183-94. doi: 10.1046/j.1360-0443.2002.00185.x. PMID 12199834
- [Background] Ghanbari B, Malakouti SK, Nojomi M, Alavi K, Khaleghparast S. Suicide Prevention and Follow-Up Services: A Narrative Review. Glob J Health Sci. 2015 Sep 28;8(5):145-53. doi: 10.5539/gjhs.v8n5p145. PMID 26652085
- [Background] Gardner, K. and P. Qualter (2009). "Reliability and validity of three screening measures of borderline personality disorder in a nonclinical population." Personality and Individual Differences 46(5-6): 636-641
- [Background] Freeman MP, Hock RS, Papakostas GI, Judge H, Cusin C, Mathew SJ, Sanacora G, Iosifescu DV, DeBattista C, Trivedi MH, Fava M. Body Mass Index as a Moderator of Treatment Response to Ketamine for Major Depressive Disorder. J Clin Psychopharmacol. 2020 May/Jun;40(3):287-292. doi: 10.1097/JCP.0000000000001209. PMID 32332464
- [Background] Forte A, Pompili M, Imbastaro B, De Luca GP, Mastrangelo M, Montalbani B, Baldessarini RJ. Effects on suicidal risk: Comparison of clozapine to other newer medicines indicated to treat schizophrenia or bipolar disorder. J Psychopharmacol. 2021 Sep;35(9):1074-1080. doi: 10.1177/02698811211029738. Epub 2021 Jul 22. PMID 34291676
- [Background] Fleischmann A, Bertolote JM, Wasserman D, De Leo D, Bolhari J, Botega NJ, De Silva D, Phillips M, Vijayakumar L, Varnik A, Schlebusch L, Thanh HT. Effectiveness of brief intervention and contact for suicide attempters: a randomized controlled trial in five countries. Bull World Health Organ. 2008 Sep;86(9):703-9. doi: 10.2471/blt.07.046995. PMID 18797646
- [Background] Feng W, Chen C, Zeng Y, Zhang B. Efficacy of single and repeated ketamine administration for suicidal ideation in adults with psychiatric disorders: A meta-analysis. Prog Neuropsychopharmacol Biol Psychiatry. 2025 Jan 10;136:111152. doi: 10.1016/j.pnpbp.2024.111152. Epub 2024 Sep 25. PMID 39332580
- [Background] Eggart V, Cordier S, Hasan A, Wagner E. Psychotropic drugs for the treatment of non-suicidal self-injury in children and adolescents: a systematic review and meta-analysis. Eur Arch Psychiatry Clin Neurosci. 2022 Dec;272(8):1559-1568. doi: 10.1007/s00406-022-01385-w. Epub 2022 Feb 16. PMID 35174411
- [Background] DeCou CR, Comtois KA, Landes SJ. Dialectical Behavior Therapy Is Effective for the Treatment of Suicidal Behavior: A Meta-Analysis. Behav Ther. 2019 Jan;50(1):60-72. doi: 10.1016/j.beth.2018.03.009. Epub 2018 Mar 22. PMID 30661567
- [Background] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Background] Danayan K, Chisamore N, Rodrigues NB, Vincenzo JDD, Meshkat S, Doyle Z, Mansur R, Phan L, Fancy F, Chau E, Tabassum A, Kratiuk K, Arekapudi A, Teopiz KM, McIntyre RS, Rosenblat JD. Real world effectiveness of repeated ketamine infusions for treatment-resistant depression with comorbid borderline personality disorder. Psychiatry Res. 2023 May;323:115133. doi: 10.1016/j.psychres.2023.115133. Epub 2023 Mar 5. PMID 36889160
- [Background] Damiano RF, Hoffmann MS, Gosmann NP, Pan PM, Miguel EC, Salum GA. Translating measurement into practice: Brazilian norms for depressive symptom assessment with the Patient Health Questionnaire (PHQ-9). Braz J Psychiatry. 2023;45(4):310-317. doi: 10.47626/1516-4446-2022-2945. Epub 2023 Mar 19. PMID 36934346
- [Background] Damiano RF, Beiram L, Damiano BBF, Hoffmann MS, Moreira-Almeida A, Ruck C, Tavares H, Brunoni AR, Miguel EC, Menezes PR, Salum GA. Associations between a Brazilian suicide awareness campaign and suicide trends from 2000 to 2019: Joinpoint and regression discontinuity analysis. J Affect Disord. 2024 Nov 15;365:459-465. doi: 10.1016/j.jad.2024.08.134. Epub 2024 Aug 24. PMID 39187205
- [Background] Cipriani A, Hawton K, Stockton S, Geddes JR. Lithium in the prevention of suicide in mood disorders: updated systematic review and meta-analysis. BMJ. 2013 Jun 27;346:f3646. doi: 10.1136/bmj.f3646. PMID 23814104
- [Background] Ciconelli, R. (1999). Tradução para a língua portuguesa e validação do questionário genérico de avaliação de qualidade de vida SF-36 (Brasil SF-36). . Revista Brasileira de Reumatologia 32: 143-150.
- [Background] Chu, C., C. R. Wilks, T. Joiner and P. M. Gutierrez (2023). "Cross-Sectional and Longitudinal Correlates of Interrupted and Aborted Suicide Attempts Among U.S. Active Duty Service Members Seeking Treatment for Suicidal Symptoms." Clinical Psychological Science 11(5): 863-878.
- [Background] Chen MH, Li CT, Lin WC, Hong CJ, Tu PC, Bai YM, Cheng CM, Su TP. Rapid inflammation modulation and antidepressant efficacy of a low-dose ketamine infusion in treatment-resistant depression: A randomized, double-blind control study. Psychiatry Res. 2018 Nov;269:207-211. doi: 10.1016/j.psychres.2018.08.078. Epub 2018 Aug 21. PMID 30153598
- [Background] Chan MK, Bhatti H, Meader N, Stockton S, Evans J, O'Connor RC, Kapur N, Kendall T. Predicting suicide following self-harm: systematic review of risk factors and risk scales. Br J Psychiatry. 2016 Oct;209(4):277-283. doi: 10.1192/bjp.bp.115.170050. Epub 2016 Jun 23. PMID 27340111
- [Background] Carter T, Walker GM, Aubeeluck A, Manning JC. Assessment tools of immediate risk of self-harm and suicide in children and young people: A scoping review. J Child Health Care. 2019 Jun;23(2):178-199. doi: 10.1177/1367493518787925. Epub 2018 Jul 29. PMID 30058359
- [Background] Carter G, Milner A, McGill K, Pirkis J, Kapur N, Spittal MJ. Predicting suicidal behaviours using clinical instruments: systematic review and meta-analysis of positive predictive values for risk scales. Br J Psychiatry. 2017 Jun;210(6):387-395. doi: 10.1192/bjp.bp.116.182717. Epub 2017 Mar 16. PMID 28302700
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Burke TA, Hamilton JL, Ammerman BA, Stange JP, Alloy LB. Suicide risk characteristics among aborted, interrupted, and actual suicide attempters. Psychiatry Res. 2016 Aug 30;242:357-364. doi: 10.1016/j.psychres.2016.05.051. Epub 2016 Jun 9. PMID 27344029
- [Background] Bryan CJ, Mintz J, Clemans TA, Leeson B, Burch TS, Williams SR, Maney E, Rudd MD. Effect of crisis response planning vs. contracts for safety on suicide risk in U.S. Army Soldiers: A randomized clinical trial. J Affect Disord. 2017 Apr 1;212:64-72. doi: 10.1016/j.jad.2017.01.028. Epub 2017 Jan 23. PMID 28142085
- [Background] Bryan CJ, Mintz J, Clemans TA, Burch TS, Leeson B, Williams S, Rudd MD. Effect of Crisis Response Planning on Patient Mood and Clinician Decision Making: A Clinical Trial With Suicidal U.S. Soldiers. Psychiatr Serv. 2018 Jan 1;69(1):108-111. doi: 10.1176/appi.ps.201700157. Epub 2017 Oct 2. PMID 28967323
- [Background] Bryan CJ, Bryan AO, Khazem LR, Aase DM, Moreno JL, Ammendola E, Bauder CR, Hiser J, Daruwala SE, Baker JC. Crisis response planning rapidly reduces suicidal ideation among U.S. military veterans receiving massed cognitive processing therapy for PTSD. J Anxiety Disord. 2024 Mar;102:102824. doi: 10.1016/j.janxdis.2023.102824. Epub 2023 Dec 21. PMID 38154445
- [Background] Bruton AM, Wesemann DG, Machingo TA, Majak G, Johnstone JM, Marshall RD. Ketamine for mood disorders, anxiety, and suicidality in children and adolescents: a systematic review. Eur Child Adolesc Psychiatry. 2025 Jan;34(1):141-157. doi: 10.1007/s00787-024-02458-y. Epub 2024 May 16. PMID 38750191
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Dartora EG, Miozzo IC, de Barba ME, Barreto SS. Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index. Sleep Med. 2011 Jan;12(1):70-5. doi: 10.1016/j.sleep.2010.04.020. Epub 2010 Dec 9. PMID 21145786
- [Background] Beck AT, Weissman A, Lester D, Trexler L. The measurement of pessimism: the hopelessness scale. J Consult Clin Psychol. 1974 Dec;42(6):861-5. doi: 10.1037/h0037562. No abstract available. PMID 4436473
- [Background] Barber ME, Marzuk PM, Leon AC, Portera L. Aborted suicide attempts: a new classification of suicidal behavior. Am J Psychiatry. 1998 Mar;155(3):385-9. doi: 10.1176/ajp.155.3.385. PMID 9501750
- [Background] Anzolin AP, Baldez DP, Montezano BB, Kapczinski F, de Abreu PB, Kauer-Sant'Anna M. Subcutaneous ketamine reduces suicide risk and improves functioning in depression: A proof-of-concept study. Psychiatry Res. 2024 Jul;337:115915. doi: 10.1016/j.psychres.2024.115915. Epub 2024 Apr 20. PMID 38688118
- [Background] Anand A, Mathew SJ, Sanacora G, Murrough JW, Goes FS, Altinay M, Aloysi AS, Asghar-Ali AA, Barnett BS, Chang LC, Collins KA, Costi S, Iqbal S, Jha MK, Krishnan K, Malone DA, Nikayin S, Nissen SE, Ostroff RB, Reti IM, Wilkinson ST, Wolski K, Hu B. Ketamine versus ECT for Nonpsychotic Treatment-Resistant Major Depression. N Engl J Med. 2023 Jun 22;388(25):2315-2325. doi: 10.1056/NEJMoa2302399. Epub 2023 May 24. PMID 37224232
- [Background] Alnefeesi Y, Chen-Li D, Krane E, Jawad MY, Rodrigues NB, Ceban F, Di Vincenzo JD, Meshkat S, Ho RCM, Gill H, Teopiz KM, Cao B, Lee Y, McIntyre RS, Rosenblat JD. Real-world effectiveness of ketamine in treatment-resistant depression: A systematic review & meta-analysis. J Psychiatr Res. 2022 Jul;151:693-709. doi: 10.1016/j.jpsychires.2022.04.037. Epub 2022 May 25. PMID 35688035
- [Background] Abbar M, Demattei C, El-Hage W, Llorca PM, Samalin L, Demaricourt P, Gaillard R, Courtet P, Vaiva G, Gorwood P, Fabbro P, Jollant F. Ketamine for the acute treatment of severe suicidal ideation: double blind, randomised placebo controlled trial. BMJ. 2022 Feb 2;376:e067194. doi: 10.1136/bmj-2021-067194. PMID 35110300